CLINICAL TRIAL: NCT03986723
Title: Evaluation of Implementation of 3D Printed Models in 3D Virtual Treatment Planning of Orthognathic Surgery
Brief Title: 3D Printed Models in 3D Virtual Treatment Planning of Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Gwen Swennen, maxillofacial surgeon, principal investigator, AZ Sint-Jan AV
Other Study IDs: 2241
Record Dates: First submitted 2019-02-14; First posted 2019-06-14 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Orthognathic Surgery
Keywords: traditional plaster model; 3D printed model; digital workflow; reliability; time efficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the shift from 2D towards 3D virtual treatment planning of orthognathic surgery, traditional plaster cast are still gold standard. The investigators aimed to compare the overall reliability and time efficiency of an digital workflow using 3D printed models, in comparison to the conventional plaster workflow.

Twenty real-life cases were planned according to both workflows and timed by a single resident.

ELIGIBILITY:
Inclusion Criteria:

* planned for orthognathic surgery
* planning by a single resident
* planning based on 3D virtual workflow

Exclusion Criteria:

* not eligible according to abovementioned criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive orthognathic cases planned with 3D virtual planning software
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
time efficiency: duration of the complete workflow, measured in seconds with a digital chronometer | preoperative
  duration of the complete workflow, measured in seconds with a digital chronometer

SECONDARY OUTCOMES:
reliability of the workflow through registration of problems, difficulties that occur | preoperative
  evaluation of the reliability of the workflow through registration of problems, difficulties that occur

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Swennen, MD PhD, Principal Investigator — AZ Sint-Lucas Brugge
Locations (1):
- AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No